CLINICAL TRIAL: NCT05896813
Title: A Prospective, Single-arm, Multicenter Clinical Study of the Combination of CMOP Regimen and Chidamide in the Treatment of Newly Diagnosed Peripheral T-cell Lymphoma
Brief Title: CMOP Regimen and Chidamide in the Treatment of Newly Diagnosed Peripheral T-cell Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DED-PTCL-K
Record Dates: First submitted 2023-06-01; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Newly Diagnosed Peripheral T-cell Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CMOP+Chi (Experimental): Cyclophosphamide: 750 mg/m2, d1; Mitoxantrone Hydrochloride Liposome: 20 mg/m2, d1; Vincristine: 1.4 g/m2, d1 (maximum dose of 2 mg), or vindesine 3 mg/m2, d1; Prednisone: 60 mg/m2, d1-d5; Chidamide:20 mg, biw. The treatment is administered every 3 weeks as a cycle and lasts for a total of 6 cycles.
  Interventions: Drug: CMOP+Chidamide

INTERVENTIONS:
Drug: CMOP+Chidamide — Cyclophosphamide: 750 mg/m2, d1; Mitoxantrone Hydrochloride Liposome: 20 mg/m2, d1; Vincristine: 1.4 g/m2, d1 (maximum dose of 2 mg), or vindesine 3 mg/m2, d1; Prednisone: 60 mg/m2, d1-d5; Chidamide:20 mg, biw. The treatment is administered every 3 weeks as a cycle and lasts for a total of 6 cycles.

SUMMARY:
Peripheral T-cell lymphoma (PTCL) is a highly heterogeneous and aggressive non-Hodgkin's lymphoma. The incidence rate of PTCL in China is much higher than the global average, and there is no unified standard treatment for initial PTCL. Currently, the CHOP regimen is widely used as first-line treatment. However, the overall response rate is still low, and effective therapies need to be explored. Epigenetics and genetics jointly determine critical features of tumors, and exploring new treatment strategies and developing targeted drugs based on deep understanding of the pathogenesis is of significant importance. The combined application of DNMT inhibitors and HDAC inhibitors has strong scientific support. The Phase II clinical study of Mitoxantrone Hydrochloride Liposome in treating relapsed or refractory PTCL achieved positive results and regulatory approval. The CMOP regimen combining Mitoxantrone Hydrochloride Liposome with Chidamide is worth exploring for initial PTCL treatment.

DETAILED DESCRIPTION:
Peripheral T-cell lymphoma (PTCL) originates from mature thymic T-cells and is a highly heterogeneous and aggressive non-Hodgkin's lymphoma (NHL). The 2016 revised WHO classification divides PTCL into 4 major categories with over 30 subtypes, including common subtypes such as anaplastic large-cell lymphoma (ALCL), ALK-positive/+ and ALK-negative/-, angioimmunoblastic T-cell lymphoma (AITL), and PTCL, not otherwise specified (PTCL-NOS) . In 2020, the estimated global incidence of new NHL patients was over 540,000, with over 90,000 cases in China. Compared with B-cell lymphomas, PTCL has a lower incidence rate, but PTCL patients' proportion in China is significantly higher than in Western countries at approximately 21% . The incidence rate of PTCL in China accounts for nearly 21% of NHL, much higher than the global average .

Currently, there is no unified standard treatment for initial PTCL. The National Comprehensive Cancer Network (NCCN) guidelines in the US and the Chinese Society of Clinical Oncology (CSCO) recommend using the CHOP regimen (cyclophosphamide, doxorubicin, vincristine, and prednisone) as first-line treatment . However, the CHOP regimen is mainly based on treatment experience with B-cell lymphomas, and more effective therapies need to be explored. Over the past few decades, research progress in both basic and clinical aspects of PTCL has been slow, with poor treatment outcomes. The overall response rate of first-line treatment is 50%-70%. Except for ALCL, ALK(+), PTCL patients receiving induction therapy are suggested to undergo autologous hematopoietic stem cell transplantation (ASCT) treatment, yet even so, the overall response rate is still low, with a poor prognosis. Except for ALCL, ALK+ patients, the five-year overall survival (OS) rate of other subtypes is less than 50% , and PTCL patients are prone to relapse , with a three-year OS probability of about 20% .

The overall treatment effect for PTCL patients is still not ideal, and their prognosis has not improved over the past few decades. Patients often relapse early, with a shorter progression-free survival (PFS) and OS. Genetic mutations, variations, and tumor occurrence and development are closely related, and the same is true for epigenetic regulation. Epigenetics and genetics jointly determine critical features of a tumor: heterogeneity, plasticity, stem cell-like properties, and immune escape. As lymphomas often have epigenetic mutations, exploring new treatment strategies and developing targeted drugs based on a deep understanding of the pathogenesis is of significant importance in improving the efficacy of PTCL treatment.

Since both highly methylated DNA and low acetylated histones can lead to a closed chromatin state by independent mechanisms, resulting in the silencing of tumor suppressor genes , the combined application of DNMT inhibitors and HDAC inhibitors has strong scientific support. Both DNMT inhibitors and HDAC inhibitors have a chemosensitizing effect. Acetylation changes the chromatin structure, plays a role in regulating epigenetics as well as in chemotherapy sensitization, while DNMT inhibitors can enhance the sensitivity of lymphoma resistant to chemotherapy. Currently, the combination of AZA+HDACi in epigenetic treatments has been explored for lymphoma treatment.

In the Phase II clinical study of Mitoxantrone Hydrochloride Liposome, 108 patients with relapsed or refractory PTCL were treated with Mitoxantrone Hydrochloride Liposome alone, achieving an objective response rate (ORR) of 41.7% (32.3%, 51.5%) and a complete response rate (CRR) of 23.1% (25/108). The median PFS was 8.5 months, and the median OS was 22.8 months. The treatment was well-tolerated and efficacious, resulting in regulatory approval for Mitoxantrone Hydrochloride Liposome in treating relapsed or refractory PTCL adult patients . Based on this, the CMOP regimen, which is based on Mitoxantrone Hydrochloride Liposome combined with Chidamide, is worth exploring for initial PTCL treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The patient understands the content of this study, voluntarily participates in the study, and signs the informed consent form (ICF);
2. Age: 18-80 years;
3. Expected survival time ≥ 3 months;
4. Histologically confirmed PTCL, one of the following subtypes:

   1. PTCL not otherwise specified (PTCL-NOS)
   2. Nodal T follicular helper (Tfh) cell lymphoma
   3. Other subtypes of PTCL that the researcher deems eligible for inclusion in the study;
5. At least one measurable or evaluable lesion that meets the Lugano2014 criteria: for lymph node lesions, the longest diameter should be >1.5 cm, and for extranodal lesions, the longest diameter should be >1.0 cm;
6. ECOG score 0-2 points;
7. Bone marrow function: neutrophil count ≥ 1.5×109/L, platelet count ≥ 75×109/L, hemoglobin ≥ 80 g/L (for patients with bone marrow involvement, the neutrophil count can be relaxed to ≥ 1.0×109/L, platelet count can be relaxed to ≥ 50×109/L, hemoglobin can be relaxed to ≥ 75 g/L);
8. Liver and kidney function: serum creatinine ≤ 1.5 times the upper limit of normal, AST and ALT ≤ 2.5 times the upper limit of normal (≤ 5 times the upper limit of normal for patients with liver involvement), and total bilirubin ≤ 1.5 times the upper limit of normal (≤ 3 times the upper limit of normal for patients with liver involvement).

Exclusion Criteria:

* 1. Hypersensitivity to any study drug or its components; 2. Uncontrollable systemic diseases (such as advanced infection, uncontrolled hypertension, diabetes, etc.); 3. One of the following applies to cardiac function and disease:

  1. Long QT syndrome or QTc interval >480 ms;
  2. Complete left bundle branch block, II or III degree atrioventricular block;
  3. Severe, uncontrolled arrhythmia requiring medication;
  4. New York Heart Association (NYHA) grade ≥ III;
  5. Left ventricular ejection fraction (LVEF) <50%;
  6. A history of acute myocardial infarction, unstable angina, severe unstable ventricular arrhythmia, or other arrhythmias or clinically significant pericardial disease requiring treatment within the six months prior to recruitment or evidence of acute ischemic or active conduction system abnormalities on the electrocardiogram; 4. Active hepatitis B or C infection (hepatitis B surface antigen positive and hepatitis B virus DNA > 1x104 copies/mL; hepatitis C virus RNA > 1x104 copies/mL); 5. Human immunodeficiency virus (HIV) infection (HIV antibody positive); 6. Previously or currently diagnosed with other malignant tumors (except for non-melanoma skin basal cell carcinoma, breast/cervical carcinoma in situ, and other malignant tumors that have not been treated and effectively controlled within the past five years); 7. Central nervous system (CNS) lymphoma or a history of CNS lymphoma; 8. Pregnant or lactating women and childbearing patients who do not want to take contraceptive measures; 9. Other situations judged by the researcher to be unsuitable for participation in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 1 year
  overall response rate

SECONDARY OUTCOMES:
CRR | 1 year
  Complete remission rate
2-year PFS | 2 years
  2-year progression-free survival
2-year OS | 2 years
  2-year overall survival
SAE | 2 years
  The frequency of serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Hematological Department, People's Hospital of Jiangsu Province, Nanjing, Jiangsu, China